CLINICAL TRIAL: NCT02849184
Title: A Multi-center, Double-blind, Randomized, Parallel Design Study to Compare the Effectiveness of Suvorexant Versus Placebo on Sleep Pressure and Circadian Rhythm in Hypertensives With Insomnia: The Super 1 Study
Brief Title: To Compare the Effectiveness of Suvorexant vs Placebo on Sleep Pressure in Hypertensives With Insomnia
Acronym: Super1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jichi Medical University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Satt Co.,Ltd (Unknown)
Responsible Party: Principal Investigator, Kazuomi Kario, Professor & Chairman, Division of Cardiovascular Medicine, Department of Medicine, Jichi Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 4305-063
Record Dates: First submitted 2016-07-21; First posted 2016-07-29 (Estimated); Results first posted 2019-08-05 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-06

CONDITIONS: Hypertension; Insomnia
MeSH Terms: conditions — Hypertension; Sleep Initiation and Maintenance Disorders | interventions — suvorexant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- suvorexant (Experimental): Suvorexant (20mg for 64 years or younger; 15mg for 65 years or older) in oral administration, once daily before bedtime; Treatment duration: 2 weeks
  Interventions: Drug: suvorexant
- placebo (Placebo Comparator): Placebo in oral administration, once daily before bedtime; Treatment duration: 2 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: suvorexant — Suvorexant (20mg for 64 years or younger; 15mg for 65 years or older) once daily before bedtime.
  Other Names: Belsomra
  Arms: suvorexant
Other: Placebo — Placebo once daily before bedtime.
  Arms: placebo

SUMMARY:
The purpose of this study is to compare the effectiveness and safety of suvorexant versus placebo on sleep pressure and circadian rhythm in hypertensives with insomnia.

DETAILED DESCRIPTION:
The study consists of a 4-week run-in period and a 2-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

[At interim registration]

Patients who meet the following criteria are eligible for the study:

1. Patients who give written consent of agreement to voluntarily participation in the clinical study
2. Age 20 years or older
3. Sex: Male or female
4. Treatment classification: Outpatient
5. Hypertensive patient who meet at least one of the following:

   * Under antihypertensive medications
   * Clinic systolic blood pressure (SBP) less than 160 mmHg
6. Patients with insomnia who meet at least one of the following:

   * Patients with any one of the following symptoms twice a week or more and at least 1 month-continuation: difficulty initiating sleep (time to sleep onset 2 hours or more longer than usual), difficulty maintaining sleep (awakening twice or more in the night), early morning awakening (awakening 2 hours or more earlier in the morning than usual), difficulty sleeping deeply (no soundly asleep feeling at the time of awakening in the morning).

     b. Patients with interference with social or occupational function due to the above insomnia symptoms

[At official registration]

Patients who meet the following criteria at the end of run-in period are eligible for the study:

1. Stable unchanged antihypertensive medication for run-in period.
2. Average morning home SBP more than 135 mmHg during 5 days before the end of run-in period.

Exclusion Criteria:

1. Patients with serious liver disease.
2. Patients with serious respiratory disease.
3. Patients with secondary hypertension
4. Patients with sleep apnea syndrome
5. Patients with history of narcolepsy or cataplexy
6. Patients with history of organic cerebral disorders
7. Patients with history of hypersensitivity to suvorexant
8. Patients received CYP3A strongly-inhibitors including itraconazole, clarithromycin and ritonavir, saquinavir, nelfinavir, indinavir, telaprevir and voriconazole at the start of the run-in period
9. Patients with average clinic SBP of 160 mmHg or more at the start of the run-in period
10. Patients received suvorexant and other hypnotic at the start of the run-in period on a regular basis
11. Patients who are breast-feeding, pregnant, possibly pregnant, or plan to become pregnant
12. Patients who are considered not to be eligible for this study by their investigator or sub-investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2017-01-17 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kazuomi Kario, MD, PhD, Principal Investigator — Jichi Medical University School of Medicine
Locations (3):
- Japan (3):
  - Takahira Internal Medicine Clinic, Fukuoka
  - Yamasaki family clinic, Hyōgo
  - Yagi hospital, Tokyo

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Suvorexant | Placebo
Started | 40 | 42
Completed | 40 | 42
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Suvorexant | Placebo | Total
Number analyzed (Participants) | 40 | 42 | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.3 (12.1) | 55.9 (9.5) | 56.6 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 13 | 24
  Male | 29 | 29 | 58
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI [Mean (Standard Deviation); unit: kg/m^2] | 25.5 (4.4) | 25.9 (3.9) | 25.7 (4.1)
Nighttime systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 137.9 (15.9) | 140.7 (18.1) | 139.4 (17.0)
Nighttime diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 80.5 (8.7) | 84.2 (10.2) | 82.4 (9.6)

OUTCOME MEASURES:

1. Primary Outcome: Change in Sleep Systolic Blood Pressure
Description: To compare the efficacy of suvorexant versus placebo on sleep systolic blood pressure (SBP) by ambulatory blood pressure monitoring (ABPM).
  Change: sleep SBP value at 2 weeks minus value at baseline
Time Frame: 2 weeks
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 40 | 42
mmHg | -1.8 (2.7) | -4.4 (2.7)

2. Secondary Outcome: Change in Morning Systolic Blood Pressure Variability
Description: To compare the efficacy of suvorexant versus placebo on morning SBP variability by ABPM Variability: SD Change: value at 2 weeks minus value at baseline
Time Frame: 2 weeks
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 40 | 42
mmHg | -0.3 (1.5) | 0.8 (1.5)

3. Secondary Outcome: Changes in the Total Sleep Time
Description: Total sleep time was assessed using a sleep diary. Value at week 2 - Value at week 0
Time Frame: 2 weeks
Measure: Mean (Standard Error); unit: hours
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 40 | 42
hours | 0.51 (0.24) | 0.43 (0.25)

4. Secondary Outcome: Changes in the Time to Sleep Onset
Description: Time to sleep onset was assessed using a sleep diary. Value at week 2 - Value at week 0
Time Frame: 2 weeks
Measure: Mean (Standard Error); unit: hours
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 40 | 42
hours | -0.23 (0.18) | -0.42 (0.15)

5. Secondary Outcome: Change in Nighttime SBP in Patients Achieved High Sleep Satisfaction
Description: nighttime BPs are measured by ambulatory blood pressure monitoring. Sleep quality is measured by self-reported sleep diary (satisfaction level of sleep) at 2 weeks.
  Patients are divided by sleep satisfaction and compared nighttime SBP change (value at 2 weeks minus value at baseline).
Time Frame: 2 weeks
Population: Patients who were satisfied with sleep as of 2 weeks
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 24 | 17
mmHg | -6.1 (3.5) | 3.1 (4.2)

6. Secondary Outcome: Change in Urinary Albumin-to-creatinine Ratio (UACR)
Description: Percentage change in UACR from baseline to 2 weeks
Time Frame: 2 weeks
Measure: Median (95% Confidence Interval); unit: percentage change
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 40 | 42
percentage change | 1.50 [-15.18 to 21.45] | -13.12 [-27.22 to 3.71]

7. Secondary Outcome: Change in Nighttime SBP in Patients Achieved Low Sleep Satisfaction
Description: nighttime BPs are measured by ambulatory blood pressure monitoring. Sleep quality is measured by self-reported sleep diary (satisfaction level of sleep) at 2weeks.
  Patients are divided by sleep satisfaction and compared nighttime SBP change (value at 2 weeks minus value at baseline).
Time Frame: 2 weeks
Population: Patients who were not satisfied with sleep as of 2 weeks
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 16 | 25
mmHg | 4.5 (3.9) | -9.5 (3.1)

8. Secondary Outcome: Change in NT-proBNP
Description: Percentage change in NT-proBNP from baseline to 2 weeks
Time Frame: 2 weeks
Measure: Median (95% Confidence Interval); unit: percentage change
Arm/Group | Suvorexant | Placebo
Number analyzed (Participants) | 40 | 42
percentage change | 3.65 [-13.90 to 24.77] | -2.80 [-19.06 to 16.72]

ADVERSE EVENTS:
Time Frame: 14 months
Arm/Group | Suvorexant | Placebo
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/42
Other Adverse Events (participants affected / at risk) | 0/40 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-10): https://cdn.clinicaltrials.gov/large-docs/84/NCT02849184/Prot_SAP_000.pdf